CLINICAL TRIAL: NCT01335854
Title: Promoting CPAP Adherence and Treatment Outcomes in Patients With Obstructive Sleep Apnea
Brief Title: Promoting Continuous Positive Airway Pressure (CPAP) Adherence
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 812091; RC2AG036592 (NIH)
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2012-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Apnea-hypopnea index; Continuous positive airway pressure; CPAP adherence
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (No Intervention): Usual care for 3 months. This consists of a phone call after one week of treatment, and clinic appointments at the sleep center following one month and three months of CPAP treatment.
- Web-Access to CPAP Data (Experimental): Usual care and web-based access to CPAP adherence data for 3 months. Participants in this group will be asked to review their CPAP use daily in the first week of treatment and as desired over the next 3 months by accessing a password protected website.
  Interventions: Behavioral: Web-based Access to CPAP Data
- Web-Access to CPAP Data & Incentive (Experimental): Usual care and web-based access to CPAP data for 3 months with financial incentives. Participants in this group will be asked to review their CPAP use daily in the first week of treatment and as desired over the next 3 months by accessing a password protected website. Financial incentive terminated after 1 week.
  Interventions: Behavioral: Web-based Access to CPAP Data with Financial Incentive

INTERVENTIONS:
Behavioral: Web-based Access to CPAP Data — Participants will have web-based access to their CPAP usage for each 24 hours of treatment. They will be asked to view this data each day during the first week of the study, and then as frequently as they choose after the first week.
  Arms: Web-Access to CPAP Data
Behavioral: Web-based Access to CPAP Data with Financial Incentive — Participants will have web-based access to their CPAP usage for each 24 hours of treatment. They will be asked to view this data each day during the first week of the the study, and then as frequently as they choose after the first week. There will be a payment of $30 during the first week for each day a participant uses CPAP for more than 4 hours the previous night and logs on to the website.
  Arms: Web-Access to CPAP Data & Incentive

SUMMARY:
The proposed research will evaluate new approaches to improving the ability of patients with obstructive sleep apnea (OSA), a breathing disorder during sleep, to use continuous positive airway pressure (CPAP), a medical device worn during sleep to treat OSA. 120 patients with newly diagnosed OSA who are being initiated on CPAP treatment will be assigned to one of 3 groups: usual care, usual care with web-based access to daily CPAP adherence, and usual care with web-based access to daily CPAP adherence and a financial incentive to use CPAP at least 4 hours/day in the first week of treatment. Measures of CPAP use, daytime sleepiness, and quality of life will evaluate whether patients provided web-based access to their daily CPAP adherence with and without financial incentive will have greater objectively measured average daily hours of CPAP use and greater improvement in functional outcomes following 3 months of treatment compared to patients receiving usual care.

The results will test the hypothesis that these behavioral interventions will improve patient adherence to CPAP during the critically important first week of treatment when many patients are deciding whether or not to use CPAP and that this initial level of adherence will be maintained over the long term despite withdrawal of the financial incentive.

DETAILED DESCRIPTION:
This is a nested clinical study in the NIH funded research project RC2AG036592, "Developing Interactive Technology to Improve Research and Health Behavior". The purpose of the research project is to create a web-based infrastructure to accelerate research in behavioral economics to improve health. Failure to adhere to medical treatments is a major cause of poor outcomes that increase health care spending. Changing unhealthful behaviors is difficult. One barrier to behavioral change is the need to provide patients with immediate, timely information about their behavior. Individual clinicians cannot maintain the frequent contact that is required, but technology and automated feedback mechanisms can keep these issues salient for patients. Internet technology is increasingly seen as an appealing tool to overcome this barrier and promote patient self-management. Recent evidence indicates that providing patients with web-based feedback of their health status may improve adherence to treatment and outcomes.

Another barrier to behavioral change is that people need frequent reinforcement of positive behavior and need that reinforcement often at the time they are making decisions (e.g., to smoke, to overeat, to take medication). Recent studies report that the use of financial incentives is an effective strategy to changing health behavior. Incentives in the form of direct payments provide valuable positive reinforcement and have been shown to change health behavior in a variety of contexts, including weight loss, medication adherence, and smoking cessation. One criticism of this approach to changing health behaviors is whether the new behavior is sustained once the financial incentive is withdrawn.

The proposed clinical study will use the web-based infrastructure that is developed by the research project to evaluate the application of these emerging new approaches in behavioral health intervention to improving CPAP adherence and consequent treatment outcomes in patients with OSA. In the proposed research study, 120 patients with newly diagnosed OSA who are being initiated on CPAP therapy will be randomized to one of three arms: 1) usual care, 2) usual care with the ability of the participant to view reports of his/her daily CPAP use on a password protected website, and 3) usual care with the ability of the participant to view reports of his/her daily CPAP use on a password protected website combined with a daily financial incentive in the first week based of hours per day of CPAP use. The proposed health behavior interventions will 1) provide patients greater access to information about their sleep disordered breathing, and 2) allow patients to become active members of their management team. Aim 1 will determine if the proposed health behavior interventions improve average daily hours of CPAP use in the first week and following 3 months of treatment. The overall hypothesis is that these behavioral interventions will improve patient adherence to CPAP during the critically important first week of treatment when many patients are deciding whether or not to use CPAP and that this initial level of adherence will be maintained over the long term despite withdrawal of the financial incentive.

Interventions designed to improve health-related behavior will only be justified if they lead to greater improvements in clinically relevant outcomes. To determine the impact of the proposed health behavior interventions to increase CPAP adherence on treatment outcomes, Aim 2 will compare measures of daytime function following 3 months of CPAP treatment across the three groups. The results of Aim 2 will demonstrate whether improvements in CPAP adherence due to web-based feedback with or without a financial incentive result in greater improvements in clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Apnea-hypopnea index (AHI) ≥ 10 events/hr on full-night in-laboratory polysomnogram (PSG) based on American Academic of Sleep Medicine (AASM) recommended scoring criteria
* Stable medical history and no change in medications, including anti-hypertensive, thyroid-related, and lipid-lowering medications, in the previous 2 months.
* Access to a telephone and the internet on all days of the week
* No regular use (> 3 times/week) of sedative or hypnotic medications in the last 2 months

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Are enrolled in other, ongoing clinical trials
* Inability to return for follow-up testing
* Previous diagnosis of another sleep disorder other than obstructive sleep apnea (OSA) (e.g., periodic limb movement disorder [≥ 15 limb movements/hr of sleep with arousal], central sleep apnea [≥ 50% of apneas on diagnostic PSG are central apneas], obesity hypoventilation syndrome, narcolepsy, or night eating syndrome
* Previous treatment with positive airway pressure, home oxygen therapy, tracheotomy, uvulopalatopharyngoplasty, or other non-nasal surgery for OSA
* Requiring oxygen or bilevel positive airway pressure for treatment of OSA
* A clinically unstable medical condition as defined by a new diagnosis or change in medical management in the previous 2 months (e.g., myocardial infarction, congestive heart failure, Cheyne-Stokes breathing, unstable angina, thyroid disease, depression or psychosis, ventricular arrhythmias, cirrhosis, surgery, or recently diagnosed cancer)
* Systolic BP > 180 mm Hg or diastolic BP > 100 mm Hg following 10 minutes at rest
* Night shift workers in situations or occupations where they regularly experience jet lag, or have irregular work schedules by history over the last 3 months
* Unable to perform tests due to inability to communicate verbally, inability to read and write; less than a 5th grade reading level; visual, hearing or cognitive impairment (e.g. previous head injury); or upper extremity motor deficit (e.g., previous stroke that prevents patient from using CPAP treatment)
* Inability to use CPAP due to claustrophobia, facial pathology, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Average daily hours of CPAP. | 3 months
  Average daily hours of CPAP use determined objectively by the mask-on time recorded by the CPAP machine.
The change in the mean total score on the Functional Outcome of Sleep Questionnaire. | 3 months
  The change in the mean total score on the Functional Outcome of Sleep Questionnaire (FOSQ-10), a validated, disease specific quality of life questionnaire.

SECONDARY OUTCOMES:
The percentage of days that the CPAP apparatus was used and the average daily hours of CPAP use on days used. | 3 months
  The percentage of days that the CPAP apparatus was used and the average daily hours of CPAP use on days used.
Total scores on the Epworth Sleepiness Scale (ESS) and the Medical Outcomes Study Short-Form-12 (SF-12). | 3 months
  Total scores on the Epworth Sleepiness Scale (ESS) and the Medical Outcomes Study Short-Form-12 (SF-12).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T Kuna, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania

REFERENCES:
- [Background] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784